CLINICAL TRIAL: NCT02750670
Title: Pilot Study of Obinutuzumab in Combination With GDP Chemotherapy for the Treatment of Relapsed or Refractory CD20+ Aggressive Non-Hodgkin Lymphoma
Brief Title: Obinutuzumab in Combination With GDP Chemotherapy in Patients With Relapsed or Refractory Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Hoffmann-La Roche (Industry); Ozmosis Research Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OZM-073; ML29885 (Other Grant/Funding Number: Roche)
Record Dates: First submitted 2016-04-15; First posted 2016-04-25 (Estimated); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Lymphoma, Non-Hodgkin's
Keywords: Lymphoma; Non-Hodgkin's; CD20+; Obinutuzumab; GDP Chemotherapy; Refractory and aggressive non-Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma | interventions — obinutuzumab; Gemcitabine; Dexamethasone; Calcium Dobesilate; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GD2P (Experimental): Obinutuzumab 1000mg by IV for 1.5-6.5 hours with Gemcitabine 1000mg/m^2 by IV for 30 minutes with dexamethasone 40mg by mouth daily and Cisplatin 75mg/m^2 by IV for 1 hour all for a duration of 3 cycles
  Interventions: Drug: Obinutuzumab; Drug: Gemcitabine; Drug: Dexamethasone; Drug: Cisplatin

INTERVENTIONS:
Drug: Obinutuzumab — Type II anti-CD20 monoclonal antibody
  Other Names: GAZYVA
Drug: Gemcitabine — Antineoplastic agent
Drug: Dexamethasone — Corticosteroid
  Other Names: Decadron
Drug: Cisplatin — Antineoplastic Agent

SUMMARY:
This is a pilot study to determine the overall survival rate and toxicities of obinutuzumab given with GDP chemotherapy for relapsed or refractory CD20+ aggressive non-Hodgkin lymphoma. Patients who have CD20+ and progressed R-CHOP therapy will be enrolled into the study. About 30 patients are planned to be enrolled from Princess Margaret Cancer Centre.

If the enrollment is very slow then additional site may be included. Patients will receive Obinutuzumab +GDP for 3 cycles intravenously. CT scan will be used to evaluate the response rate after cycle 2 and PET-CT will be used after cycle 3. Responders (complete metabolic response, partial metabolic response) should proceed to autologous stem cell transplant (ASCT). Patients who have progressed after three cycles or less are to have their protocol treatment discontinued, with subsequent treatment at investigator discretion. Patients will be followed up to 24 months from transplant done or last chemo. Mandatory tissue submission and optional tissue and blood submission are required for the correlative component of this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologic diagnosis for one of the following histologies according to the World Health Organization: documented at initial diagnosis or at relapse:

   * Diffuse large cell lymphoma, B-cell (includes primary mediastinal B-cell lymphoma, T-cell rich B-cell lymphoma);
   * Previous indolent lymphoma (follicular lymphoma, marginal zone lymphoma, including extranodal MALT lymphoma, lymphoplasmacytoid lymphoma) with transformation to diffuse large B-cell lymphoma at relapse (biopsy proof of transformation is mandatory);
   * Follicular lymphoma grade 3B;
   * Biopsy proof of disease at initial diagnosis is mandatory. A biopsy at relapse is mandatory. A histological diagnosis (core or excisional biopsy) is strongly encouraged; a cytological diagnosis is acceptable only in the event that tissue cannot be obtained.

   Patients must be CD20+ in order to be eligible for the study.
2. Clinically and/or radiologically measurable disease (1 site bidimensionally measurable). Measurements/ evaluations must be done within 28 days prior to registration.

   Baseline FDG-PET scan, if available, must be positive (known FDG-avid lymphoma)
3. Patient must have had at least one previous regimen of therapy for their disease. Patients must have relapsed or progressed after R-CHOP chemotherapy or equivalent.
4. Patient age is ≥16 years. Patients older than 70 years of age are not recommended for this study. (Note that the lower age limit at each centre will be determined by that centre's policy regarding the age at which an individual may sign his or her own consent.)
5. ECOG performance status of 0, 1, 2 or 3.
6. Patient must be considered fit for intensive chemotherapy and ASCT and an appropriate candidate to receive salvage chemotherapy and ASCT.
7. Laboratory Requirements: (must be done within 14 days of registration)

   Hematology:
   * Granulocytes (AGC) > 1.0 x 109/L (independent of growth factor support)
   * Platelets > 100 x 109/L (50 x 109/L if bone marrow involvement by lymphoma, independent of transfusion support)

   Biochemistry:
   * AST and ALT < 3x ULN
   * Serum total bilirubin < 1.5x ULN (≤ 5x ULN if Gilberts Disease)
   * Serum Creatinine < 1.5x ULN (or estimated GFR of ≥40 mL/min/1.73m2 using Cockcroft Gault formula)
   * International normalized ratio (INR) > 1.5 × the ULN in the absence of therapeutic anticoagulation
   * Partial thromboplastin time (PTT) or activated partial thromboplastin time (aPTT)
   * > 1.5 × the ULN in the absence of a lupus anticoagulant
8. A Women of childbearing potential (WOCBP) is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) and is not postmenopausal. Menopause is defined as 12 months of amenorrhea in a woman over age 45 years in the absence of other biological or physiological causes. Women of child bearing potential (who are heterosexually active) and men (who are sexually active with WOCBP), must be practicing a highly effective method of birth control (Pearl Index <1) such as oral contraceptives, intrauterine device, sexual abstinence or barrier method of contraception in conjunction with spermicidal jelly during study treatment and in female patients for 18 months after end of antibody treatment Men must agree to not donate sperm during and after the study. These restrictions apply for 18 months after the last dose of study drug.

   Women of childbearing potential must have a pregnancy test taken (either by serum beta-human chorionic gonadotropin [β-hCG]) or urine) and proven negative within 14 days prior to registration.

   Women who are pregnant or breastfeeding are ineligible for this study.
9. Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each patient must sign a consent form prior to enrollment in the trial to document their willingness to participate.
10. Patients must be accessible for treatment and follow-up. Patients randomized on this trial must be treated and followed at the participating centre. Investigators must assure themselves the patients randomized on this trial will be available for complete documentation of the treatment, response assessment, adverse events, and follow-up.
11. Protocol treatment is to begin within 5 working days of patient registration

Exclusion Criteria:

1. Patients who have been previously treated with obinutuzumab.
2. Life expectancy < 90 days
3. Patients with a history of other malignancies, except: adequately treated non-melanoma skin cancer and superficial bladder cancer, curatively treated in-situ cancer of the cervix or breast, or localized excised prostate cancer, other solid tumors curatively treated with no evidence of disease for > 5 years.
4. Active and uncontrolled central nervous system involvement, meningeal or parenchymal. Patients with CNS disease at initial presentation and who are in a CNS CR at the time of relapse are eligible. MRI scanning and / or lumbar puncture should be performed if there is clinical suspicion of active CNS disease.
5. Patients with symptoms suggestive of Progressive Multifocal Leukoencephalopathy (PML).
6. Major surgery performed within 4 weeks prior to registration.
7. Known history of human immunodeficiency virus (HIV), active Hepatitis C Virus infection, active Hepatitis B Virus infection or any uncontrolled active systemic infection requiring intravenous (IV) antibiotics. Patients with positive hepatitis B serology are defined as positive Hepatitis B surface antigen (HBsAg) or core antibody (anti-HBc). These patients should consult liver disease experts before start of treatment and should be monitored and managed following local medical standards to prevent hepatitis reactivation. Patients with Hepatitis B serology suggestive of infection are eligible if they are HBV DNA negative and concurrently treated with anti-viral therapy. Patients with a past history of hepatitis C who have eradicated the virus (defined as negative PCR for HCV RNA) are eligible.
8. Patients who have been vaccinated with live, attenuated vaccines within 4 weeks prior to registration.
9. Known history of stroke or intracranial hemorrhage within 6 months prior to registration.
10. Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of Screening, or any Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification.
11. Any serious active disease or co-morbid medical condition, including psychiatric illness, judged by the local investigator to preclude safe administration of the planned protocol treatment or required follow-up.
12. Any other serious intercurrent illness, life threatening condition, organ system dysfunction, or medical condition judged by the local investigator to compromise the subject's safety, preclude safe administration of the planned protocol treatment or required follow-up, including (for example):

    * Active, uncontrolled bacterial, fungal, or viral infection, history of chronic or recurrent infection
    * Clinically significant cardiac dysfunction or cardiovascular disease.
13. Patients are not eligible if they have a known hypersensitivity to the study drugs or their component, or a history of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies, or a known sensitivity or allergy to murine products

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2020-09-09 (Actual); Study Completion 2021-02-09 (Actual)

PRIMARY OUTCOMES:
The overall response rate (ORR) of G2DP by investigator assessment based on conventional CT imaging. | 42 days

SECONDARY OUTCOMES:
The ORR rate by central review of conventional CT imaging after 2 cycles of G2DP | 42 days
The Complete Response (CR) rate by FDG-PET scan | Post 63 days
The rate of successfully proceeding to autologous stem cell transplant (ASCT) | Post 63 days
Progression Free Survival (PFS) post ASCT (in transplanted patients) or after protocol discontinuation (in patients not transplanted). | Up to 2 years
The percentage of patients requiring dose reduction for hematologic toxicity. | Up to 63 days
Correlative studies on patient specimens markers of disease response (in tumor and blood/plasma) as well as to identify blood/plasma markers that provide additional discriminative information to FDG-PET scans | Up to 2 years
The Complete Response (CR) rate by central review of conventional CT imaging after 2 cycles of G2DP | 42 days
Overall Survival (OS) post ASCT (in transplanted patients) or after protocol discontinuation (in patients not transplanted). | Up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada